CLINICAL TRIAL: NCT03188341
Title: The Reasons of Repolarization Disturbances Disclosure in Vascular Surgery
Brief Title: Cardiac Complication After Vascular Surgery
Acronym: CCVS
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Jowita Biernawska, MD PhD, Pomeranian Medical University Szczecin
Other Study IDs: PomeranianMU
Record Dates: First submitted 2017-06-08; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Aortic Aneurysm, Abdominal; Ventricular Arrythmia; Peripheral Arterial Disease; Cardiac Complication
Keywords: vascular surgery; repolarization disturbances; cardiac complications; high risk patient; high risk procedure
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Peripheral Arterial Disease | interventions — Vascular Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Metabolic monitoring consisted of electrolytes and arterial blood gas analysis prior to anesthesia induction and at the end of the procedure.
  Blood was drawn into anticoagulant for genetic studies. Genomic DNA was isolated from peripheral blood leukocytes to investigate rs203462 AKAP10 polymorphism in the study population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- vascular surgery patients: * clinically concealed repolarization disturbances during vascular surgery procedure
  * clinically disclosed cardiac complications during and after vascular surgery procedure
  Interventions: Other: vascular surgery procedure

INTERVENTIONS:
Other: vascular surgery procedure — * an elective "open" vascular surgery procedure
  * ECG Holter recording during the procedure and 24 hours after operation (continuous electrocardiographic tracing (digital Holter ECG monitor)

SUMMARY:
The vascular surgery is a highest risk procedure when considering postoperative complications associated with the cardiovascular system. The leading clinical presentation is acute hemodynamic decompensation. However, one of the possible pathomechanisms might be repolarization disturbances. Many of perioperative risk factors of cardiac complications are modifiable. The identification may help in the global perioperative risk reduction.

Aim: The aim of the study was an identification of the factors which may release clinically overt repolarization disturbances.

Methods: The study group consisted of 100 patients, diagnosed with abdominal subrenal aortic aneurysms or peripheral arterial disease scheduled for an elective "open" vascular surgery procedure. The authors investigated whether age, gender, comorbidities or some perioperative factors (including hemodynamic, metabolic or genetic) were related to the occurrence of clinically concealed repolarization disturbances or clinically disclosed cardiac complications in postoperative time up to 30 day and one year after vascular surgery procedure.

DETAILED DESCRIPTION:
Vascular surgery is thought as the highest risk procedure in the context of cardiac complications. The range may include acute coronary syndrome, acute circulatory failure, severe arrhythmias, syncope and sudden cardiac death. The patient population is considered as a high risk, too. Popular calculators used for risk stratifications are based on preoperative patient's history and some general laboratory results. However, general status of the patient changes dynamically during vascular procedures leading to acquired increased risk. For this reason, sole preoperative risk prediction based on standard calculators is unsuitable and suboptimal. Advanced monitoring systems may record some temporary disturbances (e.g. ventricular repolarization disturbances), which may be asymptomatic. The clinical significance in postoperative risk prediction of such observations remains undefined. On the other hand, many of perioperative cardiac complications are caused by modifiable factors. The identification may help in the global perioperative risk reduction.

ELIGIBILITY:
Inclusion Criteria:

* adult patients diagnosed with abdominal subrenal aortic aneurysms or peripheral arterial disease scheduled for an elective "open" vascular surgery procedure

Exclusion Criteria:

* heart stimulation,
* atrioventricular and intraventricular conduction defects,
* atrial fibrillation recorded before of the study,
* antiarrhythmic drug treatment (except beta-blockers),
* unoptimal patient general status (uncontrolled diabetes, active infection)
* reoperation
* emergency operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with abdominal subrenal aortic aneurysms or peripheral arterial disease scheduled for an elective "open" vascular surgery procedure. The study was conducted by the team from Department of Anaesthesiology, Intensive Care and Acute Poisoning of the tertiary teaching hospital at the Pomeranian Medical University in Szczecin, Poland.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
cardiac complications | up to 30 days after vascular procedure
  cardiac complications according to European Society of Cardiology

SECONDARY OUTCOMES:
cardiac complications | during surgical procedure
  cardiac complications according to European Society of Cardiology
cardiac complications | one year
  cardiac complications according to European Society of Cardiology

CONTACTS AND LOCATIONS:
Overall Officials: Jowita Biernawska, MD, PhD, Principal Investigator — Department of Anaesthesiology and Intensive Care of the Pomeranian Medical University in Szczecin, Poland.

IPD SHARING:
Plan to Share IPD: No